CLINICAL TRIAL: NCT03932019
Title: A Randomized, Double-blind, Placebo-controled, Multi-center Phase II Clinical Trial for Evaluation of the Efficacy and Safety of Jitongning Tablet in Patients With Active Axial Spondyloarthritis(SpA)
Brief Title: Study of Jitongning Tablet to Treat Spondyloarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-JTNP-01
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Spondyloarthritis
Keywords: Jitongning Tablet, Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — jitongning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jitongning tablet High dose group (Experimental): Jitongning tablet,3tablets,bid,po
  Interventions: Drug: Jitongning tablet(High-dose )
- Jitongning tablet Low dose group (Experimental): Jitongning tablet,2tablets,bid,po Jitongning tablet placebo,1tablet,bid,po
  Interventions: Drug: Jitongning tablet(Low-dose )
- Placebo Comparator controlled group (Placebo Comparator): Placebo Comparator: Jitongning tablet placebo,3tablets,bid,po
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jitongning tablet(High-dose ) — Jitongning tablet,3tablets,bid,treat 12 weeks
  Other Names: Jitongning tablet,3tablets
  Arms: Jitongning tablet High dose group
Drug: Jitongning tablet(Low-dose ) — Jitongning tablet,2tablets,bid,treat 12 weeks Jitongning tablet placebo,1tablet,bid,treat 12 weeks
  Other Names: Jitongning tablet,2tablets,Jitongning tablet placebo,1tablet,
  Arms: Jitongning tablet Low dose group
Drug: Placebo — Jitongning tablet placebo,3tablets,bid,treat 12 weeks
  Other Names: Jitongning tablet placebo,3tablets
  Arms: Placebo Comparator controlled group

SUMMARY:
This study is to investigate the efficacy and safety of Jitongning Tablet in improving joint function and pain symptoms in active axial spondyloarthritis (SpA) patients and to explore the optimal dosage.

DETAILED DESCRIPTION:
Jitongning Tablet is a kind of traditional Chinese medicine(TCM), consists of Cortex Eucommiae, Duhuo(Radix Angelicae Pubescentis), Zhichuanwu(Radix Aconiti) , Rhizoma Corydalis, Radix Paeoniae Rubra, Radix Puerariae and Radix Glycyrrhizae. This study is being conducted to evaluate the efficacy and safety of Jitongning Tablet in patients with active axial spondyloarthritis (SpA) (Syndrome Of Kidney Yang Deficiency and Biood Stasis Stagnation), when compared with placebo and to explore the optimal dosage.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 65 years old (including 18 and 65) ;
* Meeting the diagnostic criteria for active axial SpA according to the the ASAS classification 2009, defined as satisfied 2 of the following:

  1. BASDAI score ≥ 4;
  2. In the assessment of pain numerical rating scale (NRS), spine pain NRS ≥ 4;
* Meeting the standard of TCM syndrome diagnosis for kidney yang deficiency and biood stasis stagnating syndrome;
* Sacroiliac arthritis of CT categories I(A)~Ⅲ(B) (including I(A) and Ⅲ(B));
* Human leukocyte antigen B27 (HLA-B27) is positive;
* C-reactive protein (CRP)/hypersensitive C-reactive protein (hsCRP) and/or erythrocyte sedimentation rate raised;
* Voluntary signing of informed consent.

Exclusion Criteria:

* Those who use NSAIDs in the first 2 weeks of randomization;
* In the first 4 weeks of randomization, take disease-modifying antirheumatic Chinese herbal medicine or Chemical drugs (such as sulfasalazine ,methotrexate, leflunomide, Chloroquine, Total glycosides of Tripterygium, Cyclophosphamide, Azathioprine, etc),opioid analgesics(Methadone, Morphine, etc.) ,systemic glucocorticoid therapy;
* In the first 3 months of randomization, take biological agents that have been used for spinal arthritis;
* Those who have undergone spinal surgery or joint surgery within 8 weeks before randomization;
* Patients who received intra-articular injection, spinal or paravertebral injection of corticosteroids within the first 6 months of randomization;
* The spine is completely stiff (fused);
* Any Other rheumatic immune system diseases or immunodeficiency syndromes such as ulcerative colitis, psoriasis, uveitis, etc.
* Those who have a fertility requirement within 6 months;
* Women during pregnancy and lactation;
* Suspected or indeed drug use, substance abuse, alcoholism;
* In the first 3 months of randomization, take the test or in progress;
* Serious cardiovascular, Liver , kidney, brain, mental, neurological disorders that affect informed consent and/or adverse event expression or observation;
* Abnormal liver function(the AST or ALT value is above the upper limit of the normal); Abnormal renal function (serum creatinine is above the upper limit of normal);
* Due to other circumstances, the investigator considered it inappropriate for the participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
ASAS 20 response | 12 weeks
  The percentage of subjects who achieved ASAS 20 response at 12th weeks

SECONDARY OUTCOMES:
BASDAI | 4 weeks,8weeks,12weeks
  the score changes of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at each visit compared to baseline.
  This instrument consists of six 10cm horizontal visual analog scales to measure severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness (both qualitative and quantitative). The final BASDAI score has a range of 0 to 10. The mean of which gives the BASDAI score (0-10). The severity of patient's symptoms from 0 (none) to 10 (most severe).
BASFI | 4 weeks,8weeks,12weeks
  the score changes of Bath Ankylosing Spondylitis Functional Index (BASFI) at each visit compared to baseline.
  This instrument consists of 8 specific questions regarding function in AS and 2 questions reflecting the patient's ability to cope with everyday life. Each question is answered on a 10 cm horizontal visual analog scale, the mean of which gives the BASFI score (0-10). The severity of patient's symptoms from 0 (none) to 10 (most severe).
Spinal pain | 4 weeks,8weeks,12weeks
  the score changes of Spinal pain at each visit compared to baseline. Spinal pain was scored as the average of two VAS questions about total spinal pain and nocturnal spinal pain. The mean of which gives the spinal pain score (0-10). The severity of patient's symptoms from 0 (none) to 10 (most severe).
PGA | 4 weeks,8weeks,12weeks
  the score changes of PGA at each visit compared to baseline. Patient global assessment was measured using a set of visual analogue scales (VAS) on which patients rated the severity of their disease from 0 (none) to 10 (most severe).
TCM syndrome scores | 4 weeks,8weeks,12weeks
  the score changes of TCM syndrome scores at each visit compared to baseline. This instrument consists of three primary symptoms: spinal pain, spinal function limited, morning stiffness and six secondary symptoms: nocturnal back pain、stabbing pain、Local cold pain、aversion to cold,preference for heat、heel pain、weakness in the lower back and knees. Four levels to measure severity of primary symptoms（0、2、4、6）and secondary symptoms（0、1、2、3）, respectively. Record the tongue and pulse conditions. The final score has a range of 0 to 100. The severity of patient's symptoms from 0 (none) to 100(most severe).The TCM syndrome effect calculated by nimodipine method. The effect of TCM syndrome from negative (worsen) to 100% (disappear).
CRP/hsCRP and ESR | 4 weeks,8weeks,12weeks
  the changes of CRP/hsCRP and ESR at each visit compared to baseline
Exposure of ibuprofen sustained release capsules | 12weeks
  Exposure of ibuprofen sustained release capsules in test group and placebo at 12th weeks.
  Exposure of ibuprofen sustained release capsules refers to the quantity of ibuprofen capsules patient actually took. The difference between the total dispensed quantity and the sum of recycling quantity and missing quantity gives the exposure of ibuprofen sustained release capsules. The exposure of ibuprofen sustained release capsules from 0 (none) to 372 (maximum).

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Study Director — Tasly Group, Co. Ltd.
Locations (11):
- China (11):
  - The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, Hefei, Anhui
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of hunan Medical University, Changsha, Hunan
  - Jiangsu Province Hospital of Integrated Traditional Chinese and Western Medicine, Nanjing, Jiangsu
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Province Hospital of Traditional Chinese Medicine, Kunming, Yunnan
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No